CLINICAL TRIAL: NCT04375202
Title: Treatment With COLchicine of Patients Affected by COVID-19: a Pilot Study
Brief Title: Colchicine in COVID-19: a Pilot Study
Acronym: COLVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient rate of patient accrual and newly available scientific evidence
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Prof Roberto Gerli, Principal Investigator, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001475-33
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: COVID; COVID-19; CORONAVIRUS; SARS-COV-2; COLCHICINE; IL-1
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine plus current care (Experimental): Colchicine 0.5 mg three times a day if weight is less than 100 kg; 1 mg twice a day if weight is more than 100 kg for 30 days or up to discharge. Reduce based on gastrointestinal symptoms appearance at discretion of the Investigator.
  Interventions: Drug: Colchicine 1 MG Oral Tablet
- Current care alone (No Intervention): Current care

INTERVENTIONS:
Drug: Colchicine 1 MG Oral Tablet — Tablets for oral administration, containing 1 mg of the active ingredient colchicine, administered 0.5 mg po every 8 hours x 30 days.
  Arms: Colchicine plus current care

SUMMARY:
This is an interventional, pilot, multicenter, randomized, open-label, phase 2 study, enrolling patients with COVID-19 disease. One-month rate of entering the critical stage (either a. Respiratory failure occurs and requires mechanical ventilation; b. Patients combined with other organ failure need ICU monitoring and treatment; c. Death) is the primary endpoint.

DETAILED DESCRIPTION:
This is an interventional, pilot, multicenter, randomized, open-label, phase 2 study, enrolling patients with COVID-19 disease. Participants will be randomized in a 1:1 ratio to receive Colchicine plus current care versus current care.

One-month rate of entering the critical stage (either a. Respiratory failure occurs and requires mechanical ventilation; b. Patients combined with other organ failure need ICU monitoring and treatment; c. Death) is the primary endpoint. Secondary objectives are trend of White blood cell count, Change of the "Sequential Organ failure Assessment" (SOFA), Rate of biochemical criterion (CK, ALT,ferritin) recovery, Rate of disease remission and safety of Colchicine.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for participation in the study
* Virological diagnosis of SARS-CoV-2 infection (real-time PCR)
* Hospitalized due to clinical/instrumental diagnosis of pneumonia
* Oxygen saturation at rest in ambient air ≤94%
* PaO2/FiO2 ratio of 350 to 200

Exclusion Criteria:

* Known hypersensitivity to colchicine or its excipients
* Severe diarrhea
* Patients who cannot take oral therapy
* Pregnant and lactating patients
* Patients with severe cardiac, renal insufficiency (creatinine clearance (CCL) <30 mL / min)
* Patients with kidney or liver damage [(AST or ALT> 5 times the normal limits in International Units (ULN)]; or are taking CYP3A4 enzyme - P glycoprotein inhibitors.
* Known other clinical condition that contraindicates colchicine and cannot be treated or solved according to the judgement of the clinician
* Neutrophils <1.000 / mmc
* Platelets <50.000 / mmc
* Bowel diverticulitis or perforation
* Patients already in ICU or requiring mechanical ventilation
* Patients receiving Tocilizumab
* Patients already enrolled in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of entering the critical stage | [1 month]
  Comply with any of the followings:
  1. Respiratory failure occurs and requires mechanical ventilation;
  2. Patients combined with other organ failure need ICU monitoring and treatment
  3. Death

SECONDARY OUTCOMES:
Trend of White blood cell count | [up to 30 days]
Change of the "Sequential Organ failure Assessment" (SOFA) | [up to 30 days]
Rate of biochemical criterion (CK, ALT, ferritin) recovery | [up to 30 days]
Rate of disease remission | [up to 30 days]
  Comply with any of the followings:
  1. No fever, cough and other symptoms;
  2. SPO2>94% or PaO2/FiO2 >350mmHg without oxygen inhalation

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Associazione Italiana Pneumologi Ospedalieri, Milan
  - Società Italiana di Reumatologia, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perricone C, Triggianese P, Bartoloni E, Cafaro G, Bonifacio AF, Bursi R, Perricone R, Gerli R. The anti-viral facet of anti-rheumatic drugs: Lessons from COVID-19. J Autoimmun. 2020 Jul;111:102468. doi: 10.1016/j.jaut.2020.102468. Epub 2020 Apr 17. PMID 32317220
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014
- See also: Related Info — https://www.aifa.gov.it/sperimentazioni-cliniche-covid-19